CLINICAL TRIAL: NCT06269939
Title: Evaluation of a Theory-Driven Manualized Approach to Improving New Learning and Memory in Healthy Aging and Mild Cognitive Impairment
Brief Title: Theory-Driven Manualized Approach to Improving New Learning and Memory in Healthy Aging and MCI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Nancy Chiaravalloti, Director, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R-1253-24
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Aging
Keywords: memory
MeSH Terms: interventions — Microscopy, Electron, Scanning Transmission

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): The experimental group will receive memory techniques training administered twice a week for four weeks (8 training sessions).
  Interventions: Behavioral: STEM
- Control group (Placebo Comparator): The control group will receive memory exercises administered twice a week for four weeks (8 sessions).
  Interventions: Behavioral: STEM

INTERVENTIONS:
Behavioral: STEM — Memory technique training

SUMMARY:
The purpose of this research study is to investigate the effectiveness of a memory enhancement technique in an aging population.

DETAILED DESCRIPTION:
Memory enhancing techniques have been incorporated into an 8-session treatment protocol, Strategy Based Training to Enhance Memory (STEM), designed to teach participants about each of the techniques, train them on how to apply the techniques in daily life and practice their application to daily life memory demanding situations. The protocol includes teaching participants over age 60 how to restructure a memory demanding situation in order to make optimal use of the techniques.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  * read and speak English fluently

Exclusion Criteria:

* prior stroke or neurological injury/disease (i.e. traumatic brain injury, Multiple Sclerosis, or Stroke).
* history of significant psychiatric illness (for example, bipolar disorder, schizophrenia, or psychosis).
* significant alcohol or drug abuse history (inpatient treatment).
* Benzodiazepines and steroid use
* Diagnosis of dementia

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Verbal Leaning task | Three points in time: pre-treatment, immediately following treatment, and 6- months after treatment is completed]
  Change in total score from Open-Trial Selective Reminding Test (OT-SRT)
Participation in Everyday life | Three points in time: pre-treatment, immediately following treatment, and 6- months after treatment is completed]
  Change in total score from Participation Assessment with Recombined Tools

SECONDARY OUTCOMES:
Functional Neuroimaging | Two points in time: pre-treatment, immediately following treatment
  Change in total scores from memory task during fMRI scan

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided